CLINICAL TRIAL: NCT00221546
Title: Influence of DHA-rich Supplement on DHA-status and Health Evolution of Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgian Society against Cystic Fibrosis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2001/220
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHA-rich supplement (Active Comparator)
  Interventions: Drug: Giving DHA-rich supplement
- Placebo (Placebo Comparator)
  Interventions: Drug: Giving DHA-rich supplement

INTERVENTIONS:
Drug: Giving DHA-rich supplement — Giving DHA-rich supplement to patients.

SUMMARY:
Investigation of the influence of giving DHA-rich supplement versus placebo on DHA-status and health evolution of patients with cystic fibrosis

DETAILED DESCRIPTION:
Investigation of the influence of giving DHA-rich supplement versus placebo on DHA-status and health evolution of patients with cystic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Delta F 508 homozygote
* Stable clinical situation

Exclusion Criteria:

-

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Clinical evolution: weight, height, pulmonary function and infection frequency before the study start and during the 2 years of the study | before the study start and during the 2 years of the study

SECONDARY OUTCOMES:
Evolution of the fatty acid profile | during the 2 years of the study
Oxidative stress status | during the 2 years of the study

CONTACTS AND LOCATIONS:
Overall Officials: Armand Christophe, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be